CLINICAL TRIAL: NCT03270514
Title: Postoperative Analgesia After Cardiac Surgery - A Double-Blind, Prospective and Randomized Comparison of Wound Infiltration With Liposomal Bupivacaine and Bupivacaine Hydrochloride
Brief Title: Comparison of Sternal Wound Infiltration With Liposomal Bupivacaine v. Bupivacaine Hydrochloride
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kathirvel Subramaniam (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor-Investigator, Kathirvel Subramaniam, Principal Investigator, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO17060305
Record Dates: First submitted 2017-08-10; First posted 2017-09-01 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenoses; Valve Regurgitation, Mitral; Valve Regurgitation, Tricuspid
Keywords: cardiac surgery; sternotomy; post-operative pain; sternal wound infiltration
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Mitral Valve Insufficiency; Tricuspid Valve Insufficiency; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care provider, investigator, and outcomes assessor are all blinded to the treatment allocation in double-blind fashion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Exparel Injectable Product (Experimental): Liposomal Bupivacaine (Exparel) Injection administered approximately 20 cc per inch of sternotomy wound. Half of subjects enrolled will be randomized to the liposomal bupivacaine (Exparel) group (~30).
  Interventions: Drug: Exparel Injectable Product
- Bupivacaine Hydrochloride (Active Comparator): Bupivacaine Injection administered approximately 20 cc per inch of sternotomy wound. Half of subjects enrolled will be randomized to the bupivacaine group (~30).
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Exparel Injectable Product — Liposomal bupivacaine 20 cc (226 mg) + Bupivacaine Hydrochloride 0.25% 40 cc (100 mg) + made up to calculated volume with normal saline solution based on the length of the incision and number of chest tubes (20 cc per tube + 20cc per inch of incision)
  Other Names: Liposomal Bupivacaine
  Arms: Exparel Injectable Product
Drug: Bupivacaine Hydrochloride — Bupivacaine 0.25% 2 mg/kg not to exceed 150 mg - made up to made up to calculated volume with normal saline solution based on the length of the incision and number of chest tubes (20 cc per tube + 20cc per inch of incision)
  Other Names: Bupivacaine
  Arms: Bupivacaine Hydrochloride

SUMMARY:
The aim of this study is to evaluate the analgesic efficacy and safety of wound infiltration with liposomal bupivacaine (LB) in patients undergoing cardiac surgery with sternotomy and cardiopulmonary bypass (CPB) and compare it with bupivacaine hydrochloride infiltration

DETAILED DESCRIPTION:
There are no studies to date on the use of LB infiltration and its analgesic efficacy in cardiac surgery done through sternotomy, even though the majority of cardiac surgeries utilize this approach. Moderate to severe pain is common in patients undergoing these surgeries and is usually inadequately treated. Other various pain treatment modalities such as opioid and neuraxial anesthesia are avoided due to potentially dangerous side effects in this cohort. The efficacy of local anesthesia techniques, such as bupivacaine, are limited due to short duration of action and increased incidence of wound infection. On the other hand, slow release liposomal bupivacaine may last up to 72 hours, indicating it's potential for more adequate analgesia compared to bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Open cardiac surgery through sternotomy approach (eg. coronary artery bypass graft, valvular heart procedures, as well as other open cardiac procedures along with coronary artery bypass)
* Surgery with the use of cardiopulmonary bypass

Exclusion Criteria:

* Minimally invasive heart surgery through thoracotomy approach
* Patient undergoing procedures under deep hypothermic circulatory arrest
* Patients with active infections such as infective endocarditis
* Emergency surgery
* Patients undergoing transplantations and ventricular assist device insertion
* Patients on any mechanical circulatory support preoperatively
* Patient's refusal
* End stage liver or renal disease
* Allergy to bupivacaine
* Patient who cannot understand the study procedure or refuse to participate
* Redo-sternotomy
* Participation in another study
* Patients with severe right or left ventricular dysfunction (EF< 25%)
* Patients requiring chronic opioids for chronic pain condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2020-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathirvel Subramaniam, MD, MPH, Principal Investigator — Associate Professor and staff Anesthesiologist
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bigeleisen PE, Goehner N. Novel approaches in pain management in cardiac surgery. Curr Opin Anaesthesiol. 2015 Feb;28(1):89-94. doi: 10.1097/ACO.0000000000000147. PMID 25500688
- [Background] Sun XL, Zhao ZH, Ma JX, Li FB, Li YJ, Meng XM, Ma XL. Continuous Local Infiltration Analgesia for Pain Control After Total Knee Arthroplasty: A Meta-analysis of Randomized Controlled Trials. Medicine (Baltimore). 2015 Nov;94(45):e2005. doi: 10.1097/MD.0000000000002005. PMID 26559294
- [Background] Tong YC, Kaye AD, Urman RD. Liposomal bupivacaine and clinical outcomes. Best Pract Res Clin Anaesthesiol. 2014 Mar;28(1):15-27. doi: 10.1016/j.bpa.2014.02.001. Epub 2014 Mar 15. PMID 24815964
- [Background] Kalogera E, Bakkum-Gamez JN, Weaver AL, Moriarty JP, Borah BJ, Langstraat CL, Jankowski CJ, Lovely JK, Cliby WA, Dowdy SC. Abdominal Incision Injection of Liposomal Bupivacaine and Opioid Use After Laparotomy for Gynecologic Malignancies. Obstet Gynecol. 2016 Nov;128(5):1009-1017. doi: 10.1097/AOG.0000000000001719. PMID 27741199
- [Background] Hutchins JL, Kesha R, Blanco F, Dunn T, Hochhalter R. Ultrasound-guided subcostal transversus abdominis plane blocks with liposomal bupivacaine vs. non-liposomal bupivacaine for postoperative pain control after laparoscopic hand-assisted donor nephrectomy: a prospective randomised observer-blinded study. Anaesthesia. 2016 Aug;71(8):930-7. doi: 10.1111/anae.13502. Epub 2016 May 30. PMID 27238859
- [Background] Hutchins J, Delaney D, Vogel RI, Ghebre RG, Downs LS Jr, Carson L, Mullany S, Teoh D, Geller MA. Ultrasound guided subcostal transversus abdominis plane (TAP) infiltration with liposomal bupivacaine for patients undergoing robotic assisted hysterectomy: A prospective randomized controlled study. Gynecol Oncol. 2015 Sep;138(3):609-13. doi: 10.1016/j.ygyno.2015.06.008. Epub 2015 Jun 6. PMID 26056753
- [Background] Beck DE, Margolin DA, Babin SF, Russo CT. Benefits of a Multimodal Regimen for Postsurgical Pain Management in Colorectal Surgery. Ochsner J. 2015 Winter;15(4):408-12. PMID 26730224
- [Background] Knudson RA, Dunlavy PW, Franko J, Raman SR, Kraemer SR. Effectiveness of Liposomal Bupivacaine in Colorectal Surgery: A Pragmatic Nonsponsored Prospective Randomized Double Blinded Trial in a Community Hospital. Dis Colon Rectum. 2016 Sep;59(9):862-9. doi: 10.1097/DCR.0000000000000648. PMID 27505115
- [Background] Ayad S, Babazade R, Elsharkawy H, Nadar V, Lokhande C, Makarova N, Khanna R, Sessler DI, Turan A. Comparison of Transversus Abdominis Plane Infiltration with Liposomal Bupivacaine versus Continuous Epidural Analgesia versus Intravenous Opioid Analgesia. PLoS One. 2016 Apr 15;11(4):e0153675. doi: 10.1371/journal.pone.0153675. eCollection 2016. PMID 27082959
- [Background] Knight RB, Walker PW, Keegan KA, Overholser SM, Baumgartner TS, Ebertowski JS 2nd, Aden JK, White MA. A Randomized Controlled Trial for Pain Control in Laparoscopic Urologic Surgery: 0.25% Bupivacaine Versus Long-Acting Liposomal Bupivacaine. J Endourol. 2015 Sep;29(9):1019-24. doi: 10.1089/end.2014.0769. Epub 2015 Jun 5. PMID 25897552
- [Background] Routman HD, Israel LR, Moor MA, Boltuch AD. Local injection of liposomal bupivacaine combined with intravenous dexamethasone reduces postoperative pain and hospital stay after shoulder arthroplasty. J Shoulder Elbow Surg. 2017 Apr;26(4):641-647. doi: 10.1016/j.jse.2016.09.033. Epub 2016 Nov 15. PMID 27856266
- [Background] Okoroha KR, Lynch JR, Keller RA, Korona J, Amato C, Rill B, Kolowich PA, Muh SJ. Liposomal bupivacaine versus interscalene nerve block for pain control after shoulder arthroplasty: a prospective randomized trial. J Shoulder Elbow Surg. 2016 Nov;25(11):1742-1748. doi: 10.1016/j.jse.2016.05.007. Epub 2016 Jul 14. PMID 27422692
- [Background] Kuang MJ, Du Y, Ma JX, He W, Fu L, Ma XL. The Efficacy of Liposomal Bupivacaine Using Periarticular Injection in Total Knee Arthroplasty: A Systematic Review and Meta-Analysis. J Arthroplasty. 2017 Apr;32(4):1395-1402. doi: 10.1016/j.arth.2016.12.025. Epub 2016 Dec 23. PMID 28082044
- [Background] Ma J, Zhang W, Yao S. Liposomal bupivacaine infiltration versus femoral nerve block for pain control in total knee arthroplasty: A systematic review and meta-analysis. Int J Surg. 2016 Dec;36(Pt A):44-55. doi: 10.1016/j.ijsu.2016.10.007. Epub 2016 Oct 11. PMID 27742564
- [Background] Yu SW, Szulc AL, Walton SL, Davidovitch RI, Bosco JA, Iorio R. Liposomal Bupivacaine as an Adjunct to Postoperative Pain Control in Total Hip Arthroplasty. J Arthroplasty. 2016 Jul;31(7):1510-5. doi: 10.1016/j.arth.2016.01.004. Epub 2016 Jan 21. PMID 26872584
- [Background] Cherian JJ, Barrington J, Elmallah RK, Chughtai M, Mistry JB, Mont MA. Liposomal Bupivacaine Suspension, Can Reduce Length of Stay and Improve Discharge Status of Patients Undergoing Total Hip Arthroplasty. Surg Technol Int. 2015 Nov;27:235-9. PMID 26680403
- [Background] Barrington JW, Olugbode O, Lovald S, Ong K, Watson H, Emerson RH Jr. Liposomal Bupivacaine: A Comparative Study of More Than 1000 Total Joint Arthroplasty Cases. Orthop Clin North Am. 2015 Oct;46(4):469-77. doi: 10.1016/j.ocl.2015.06.003. Epub 2015 Aug 6. PMID 26410636
- [Background] Barrington JW, Halaszynski TM, Sinatra RS, Expert Working Group On Anesthesia And Orthopaedics Critical Issues In Hip And Knee Replacement Arthroplasty FT. Perioperative pain management in hip and knee replacement surgery. Am J Orthop (Belle Mead NJ). 2014 Apr;43(4 Suppl):S1-S16. PMID 24911869
- [Background] Kim J, Burke SM, Kryzanski JT, Roberts RJ, Roguski M, Qu E, Hwang SW, Liu PP, Desilier A, Riesenburger RI. The Role of Liposomal Bupivacaine in Reduction of Postoperative Pain After Transforaminal Lumbar Interbody Fusion: A Clinical Study. World Neurosurg. 2016 Jul;91:460-7. doi: 10.1016/j.wneu.2016.04.058. Epub 2016 Apr 22. PMID 27113396
- [Background] Grieff AN, Ghobrial GM, Jallo J. Use of liposomal bupivacaine in the postoperative management of posterior spinal decompression. J Neurosurg Spine. 2016 Jul;25(1):88-93. doi: 10.3171/2015.11.SPINE15957. Epub 2016 Mar 4. PMID 26943250
- [Background] Abdelsattar JM, Boughey JC, Fahy AS, Jakub JW, Farley DR, Hieken TJ, Degnim AC, Goede W, Mohan AT, Harmsen WS, Niesen AD, Tran NV, Bakri K, Jacobson SR, Lemaine V, Saint-Cyr M. Comparative Study of Liposomal Bupivacaine Versus Paravertebral Block for Pain Control Following Mastectomy with Immediate Tissue Expander Reconstruction. Ann Surg Oncol. 2016 Feb;23(2):465-70. doi: 10.1245/s10434-015-4833-4. Epub 2015 Aug 26. PMID 26307232
- [Background] Smoot JD, Bergese SD, Onel E, Williams HT, Hedden W. The efficacy and safety of DepoFoam bupivacaine in patients undergoing bilateral, cosmetic, submuscular augmentation mammaplasty: a randomized, double-blind, active-control study. Aesthet Surg J. 2012 Jan;32(1):69-76. doi: 10.1177/1090820X11430831. Epub 2011 Dec 16. PMID 22179931
- [Background] Oppenheimer AJ, Fiala TGS, Oppenheimer DC. Direct Transversus Abdominis Plane Blocks With Exparel During Abdominoplasty. Ann Plast Surg. 2016 Nov;77(5):499-500. doi: 10.1097/SAP.0000000000000659. PMID 26545224
- [Background] Morales R Jr, Mentz H 3rd, Newall G, Patronella C, Masters O 3rd. Use of abdominal field block injections with liposomal bupivicaine to control postoperative pain after abdominoplasty. Aesthet Surg J. 2013 Nov 1;33(8):1148-53. doi: 10.1177/1090820X13510720. Epub 2013 Nov 8. PMID 24214950
- [Background] Golf M, Daniels SE, Onel E. A phase 3, randomized, placebo-controlled trial of DepoFoam(R) bupivacaine (extended-release bupivacaine local analgesic) in bunionectomy. Adv Ther. 2011 Sep;28(9):776-88. doi: 10.1007/s12325-011-0052-y. Epub 2011 Aug 12. PMID 21842428
- [Background] Vyas KS, Rajendran S, Morrison SD, Shakir A, Mardini S, Lemaine V, Nahabedian MY, Baker SB, Rinker BD, Vasconez HC. Systematic Review of Liposomal Bupivacaine (Exparel) for Postoperative Analgesia. Plast Reconstr Surg. 2016 Oct;138(4):748e-756e. doi: 10.1097/PRS.0000000000002547. PMID 27673545
- [Background] Khalil KG, Boutrous ML, Irani AD, Miller CC 3rd, Pawelek TR, Estrera AL, Safi HJ. Operative Intercostal Nerve Blocks With Long-Acting Bupivacaine Liposome for Pain Control After Thoracotomy. Ann Thorac Surg. 2015 Dec;100(6):2013-8. doi: 10.1016/j.athoracsur.2015.08.017. Epub 2015 Oct 24. PMID 26507422
- [Background] Balkhy HH, Arnsdorf S, Krienbring D, Urban J. Liposome Bupivacaine for Postsurgical Analgesia in Patients Undergoing Robotically Assisted Cardiac Surgery. Innovations (Phila). 2015 Nov-Dec;10(6):416-9. doi: 10.1097/IMI.0000000000000190. PMID 26633002

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [60 to 72] | 65 [60 to 72] | 65.5 [60 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 24 | 26 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 28 | 57
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 26 | 28 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 32 [29.4 to 34] | 31.3 [28.7 to 33.1] | 31.7 [29.2 to 33.6]
Diabetes mellitus [Count of Participants; unit: Participants] | 15 | 14 | 29
Hypertension [Count of Participants; unit: Participants] | 27 | 28 | 55
Congestive heart failure [Count of Participants; unit: Participants] | 5 | 5 | 10
Tobacco use [Count of Participants; unit: Participants] | 12 | 15 | 27
Chronic lung disease [Count of Participants; unit: Participants]
  Mild or no disease | 26 | 31 | 57
  Severe | 2 | 0 | 2
  Unknown | 1 | 0 | 1
Peripheral vascular disease [Count of Participants; unit: Participants] | 2 | 2 | 4
Cerebrovascular disease [Count of Participants; unit: Participants] | 1 | 2 | 3
Preoperative hospitalization [Count of Participants; unit: Participants] | 17 | 15 | 32
Hematocrit [Median (Inter-Quartile Range); unit: Percentage Hematocrit] | 40.7 [36.6 to 43.4] | 41.8 [38.6 to 44.3] | 41.5 [37.9 to 43.9]
Serum creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 1.0 [0.85 to 1.3] | 1.0 [0.9 to 1.2] | 1.0 [0.9 to 1.2]
Total albumin [Median (Inter-Quartile Range); unit: g/dL] | 4 [3.8 to 4.4] | 4.1 [3.8 to 4.3] | 4 [3.8 to 4.3]
Total bilirubin [Median (Inter-Quartile Range); unit: mg/dL] | 0.6 [0.4 to 0.8] | 0.6 [0.4 to 0.8] | 0.6 [0.4 to 0.8]
Last hemoglobin A1C [Median (Inter-Quartile Range); unit: percentage A1C] | 6.2 [5.6 to 7.2] | 6.0 [5.7 to 7.5] | 6.1 [5.7 to 7.2]
Society of thoracic surgeons predicted mortality risk [Median (Inter-Quartile Range); unit: percentage of mortality risk] — The Society of Thoracic Surgeons' risk models predict the risk of operative mortality. The risk is reported as percentage values ranging from 0-100%, where higher percentages reflect greater risk of mortality
  percentage of mortality risk | 0.009 [0.005 to 0.013] | 0.007 [0.005 to 0.013] | 0.008 [0.005 to 0.013]
Left ventricular ejection fraction [Median (Inter-Quartile Range); unit: percent ejection fraction] | 57.5 [46.5 to 58] | 58 [45 to 62] | 58 [47.3 to 60]
Angiotensin converting enzyme inhibitor/angiotensin receptor blocker use [Count of Participants; unit: Participants] — Within 48 hours preoperatively
  Participants | 6 | 4 | 10
Betablockers within 2 weeks preoperatively [Count of Participants; unit: Participants] | 22 | 18 | 40
Aspirin within 5 days preoperatively [Count of Participants; unit: Participants] | 25 | 30 | 55
Lipid lowering drugs within 24 hours preoperatively [Count of Participants; unit: Participants] | 19 | 25 | 44
Procedure [Count of Participants; unit: Participants]
  Coronary artery bypass graft | 25 | 25 | 50
  Valve procedure | 1 | 3 | 4
  Combined coronary artery bypass graft & valve procedure | 3 | 3 | 6
Duration of cardiopulmonary bypass [Median (Inter-Quartile Range); unit: minutes] | 128 [99.5 to 157] | 134 [114 to 177] | 129 [112 to 163]
Lowest body temperature on bypass [Median (Inter-Quartile Range); unit: degrees Celcius] | 34.2 [33 to 35.1] | 33.8 [32.6 to 34.8] | 34 [33 to 35]
Duration of surgery [Median (Inter-Quartile Range); unit: minutes] | 305 [279 to 385] | 335 [267 to 411] | 329 [271 to 401]

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Intensity
Description: Postoperative pain scores evaluated by numeric rating scale or (NRS) where 0- no pain and 10- worst pain, at rest and at movement
Time Frame: NRS scores will be evaluated every 4 hours until 24 hours post-operatively, every 8 hours until 48 hours post-operatively, and every 12 hours for 72 hours post-operatively
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
score on a scale
  4hrs. at rest | 4.7482 [0 to 10] | 5.03 [0 to 10]
  4hrs. with movement | 5.75 [0 to 10] | 6.64 [0 to 10]
  8hrs. at rest | 4.7262 [0 to 10] | 4.996 [0 to 10]
  8hrs. with movement | 5.74 [0 to 10] | 6.6 [0 to 10]
  12hrs. at rest | 4.7042 [0 to 10] | 4.962 [0 to 10]
  12hrs. with movement | 5.73 [0 to 10] | 6.56 [0 to 10]
  16hrs. at rest | 4.6822 [0 to 10] | 4.928 [0 to 10]
  16hrs. with movement | 5.72 [0 to 10] | 6.52 [0 to 10]
  20hrs. at rest | 4.6602 [0 to 10] | 4.894 [0 to 10]
  20hrs. with movement | 5.71 [0 to 10] | 6.48 [0 to 10]
  24hrs. at rest | 4.6382 [0 to 10] | 4.86 [0 to 10]
  24hrs. with movement | 5.7 [0 to 10] | 6.44 [0 to 10]
  32hrs. at rest | 4.5942 [0 to 10] | 4.792 [0 to 10]
  32hrs. with movement | 5.68 [0 to 10] | 6.32 [0 to 10]
  40hrs. at rest | 4.5282 [0 to 10] | 4.724 [0 to 10]
  40hrs. with movement | 5.66 [0 to 10] | 6.24 [0 to 10]
  48hrs. at rest | 4.4622 [0 to 10] | 4.656 [0 to 10]
  48hrs. with movement | 5.64 [0 to 10] | 6.16 [0 to 10]
  60hrs. at rest | 4.3742 [0 to 10] | 4.554 [0 to 10]
  60hrs. with movement | 5.61 [0 to 10] | 6.04 [0 to 10]
  72hrs. at rest | 4.2862 [0 to 10] | 4.452 [0 to 10]
  72hrs. with movement | 5.58 [0 to 10] | 5.92 [0 to 10]

2. Primary Outcome: Total Narcotic Consumption
Description: All narcotics administered in the first 0-8, 8-24, 24-48, and 48-72 hours and the total narcotics administered in the 0-72 hours postoperative period(PCA narcotics, nurse-administered IV narcotics, and oral narcotics). All narcotics will be converted to total IV morphine equivalent for comparison between two groups.
Time Frame: 0-72 hours post-operative period
Measure: Median (Inter-Quartile Range); unit: oral morphine equivalents in mg
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
oral morphine equivalents in mg
  0-8 hours | 15 [7.5 to 30] | 10 [0 to 19]
  8-24 hours | 45 [30 to 60] | 34.5 [15 to 52.5]
  24-48 hours | 45 [10 to 75] | 45 [12 to 67.5]
  48-72 hours | 15 [2.5 to 53] | 26.5 [5 to 45]
  0-72 hours | 139 [73 to 212] | 105 [54.5 to 188]

3. Secondary Outcome: Time to Extubation
Description: The time it takes until the patient is extubated post-operatively will be measured
Time Frame: From the end of surgery until the patient is extubated up to 72 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
hours | 3.85 [2.65 to 8.17] | 3.47 [2.49 to 9.58]

4. Secondary Outcome: Patient Time to Mobilization
Description: The time it takes until patient ambulates will be measured
Time Frame: From time of end of surgery to time of mobilization up to 72 hours or discharge, *assessed up to 120 hours*
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
hours | 42 [19 to 51] | 45 [33 to 78]

5. Secondary Outcome: Patient Time to Out of Bed to Chair
Description: The time it takes until the patient advances from bedrest to out of bed (OOB) to chair will be measured
Time Frame: From time of end of surgery to time of mobilization up to 72 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
hours | 16 [11 to 19] | 16 [8 to 20]

6. Secondary Outcome: Patient Time to Oral Intake
Description: The time it takes until the patient is able to/medically cleared to consume food or liquid will be measured
Time Frame: From time of end of surgery to time of oral intake up to 72 hours post-operatively or until hospital discharge
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
hours | 7 [5 to 18] | 5.6 [4.0 to 18]

7. Secondary Outcome: Non-invasive Ventilation (NIV) Requirement
Description: Episodes of NIV such as upper airway masks or similar devices will be quantified
Time Frame: From time of end of surgery to 72 hours post-operatively or until hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
Participants | 6 | 5

8. Secondary Outcome: Re-intubation
Description: Instances of re-intubation will be recorded
Time Frame: From time of end of surgery to patient discharge up to one week
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
Participants | 3 | 3

9. Secondary Outcome: Use of Incentive Spirometry
Description: Frequency of incentive spirometry will be measured
Time Frame: From time of end of surgery to 72 hours post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
Participants | 29 | 31

10. Secondary Outcome: Post-operative Nausea and Vomiting
Description: Whether a patient experiences at least one episode of nausea and emesis will be measured
Time Frame: From time of end of surgery to 72 hours post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
Participants | 3 | 9

11. Secondary Outcome: Major Organ Dysfunction
Description: Organ systems such as cardiac, renal, respiratory, and nervous system failure/dysfunction in accordance with the Society of Thoracic Surgeon's database will be noted
Time Frame: From date of surgery assessed up to 30 day post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
Participants
  Pneumonia | 1 | 0
  Renal failure / hemodialysis | 1 | 1
  Cardiac arrest | 0 | 1
  Atrial fibrillation | 7 | 15
  No major organ dysfunction | 20 | 14

12. Secondary Outcome: Length of Hospital and ICU Stay
Description: Length of both hospital and ICU stay will be measured
Time Frame: From date of surgery assessed up to 30 day post-operatively
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
days
  Length of ICU stay | 1.51 [1.08 to 2.11] | 1.71 [1.11 to 2.97]
  Length of postoperative hospital stay | 7 [5.5 to 8] | 6 [5 to 7.3]

13. Secondary Outcome: Hospital Readmission
Description: Readmission to hospital will be noted
Time Frame: From end of surgery assessed up to 30 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
Participants | 3 | 3

14. Secondary Outcome: Mortality
Description: Mortality will be noted at specific timepoints
Time Frame: From end of surgery assessed up to 30 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
Participants | 0 | 1

15. Other Pre Specified Outcome: Delirium
Description: Patients will be assessed for delirium using the Intensive Care Delirium Screening Checklist (ICDSC)
Time Frame: Assessment will be administered at 48 hours post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
Participants
  No delirium at 48 hours postoperatively | 18 | 18
  Delirium at 48 hours postoperatively | 7 | 7
  No delirium assessment conducted at 48 hours postoperatively | 4 | 6

16. Other Pre Specified Outcome: Delirium
Description: Patients will be assessed for delirium using the Intensive Care Delirium Screening Checklist (ICDSC)
Time Frame: Assessment will be administered at 72 hours post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
Participants
  No delirium at 72 hours postoperatively | 22 | 21
  Subsyndromal delirium at 72 hours postoperatively | 4 | 3
  Delirium at 72 hours postoperatively | 1 | 0
  No delirium assessment conducted at 72 hours postoperatively | 2 | 7

17. Other Pre Specified Outcome: Patient Satisfaction
Description: Patient will give an assessment regarding pain management on a scale of 0 - 10 with 0 indicating the lowest satisfaction with pain management and 10 indicating the highest satisfaction with pain management
Time Frame: Given at the time of discharge up to 30 days post-operatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
score on a scale | 10 [8 to 10] | 10 [9 to 10]

18. Other Pre Specified Outcome: Chronic Pain Assessment
Description: Subjects will be asked the two following questions: "Are you currently experiencing pain?" as well as "Are you experiencing moderate to severe pain?" with moderate to severe indicated as a pain score of 4-10 on 0 to 10 scale, with 0 being no pain at all and 10 being the worst pain imaginable.
Time Frame: 6 months after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
Participants
  Any pain at 6 months | 9 | 14
  Moderate to severe pain at 6 months | 3 | 6
  No pain at 6 months | 17 | 11

19. Other Pre Specified Outcome: Chronic Pain Assessment
Description: as for outcome 18
Time Frame: 12 months after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
Participants
  Any pain at 12 months | 7 | 12
  Moderate to severe pain at 12 months | 4 | 6
  No pain at 12 months | 18 | 13

20. Other Pre Specified Outcome: Serum Cortisol Levels
Description: Stress response suppression as a result of treatment will be evaluated by comparing hormone levels between the groups. Serum cortisol levels will be taken to measure this.
Time Frame: Measured 8, 48, and 72 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: µg/dL
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
Number analyzed (Participants) | 29 | 31
µg/dL
  8 hours postoperatively | 30 [23 to 40] | 36.5 [27 to 49]
  48 hours postoperatively | 15 [11 to 20] | 19 [14 to 24]
  72 hours postoperatively | 16 [11 to 18] | 17 [13 to 22]

ADVERSE EVENTS:
Time Frame: from the time of consent, adverse events were monitored for 30 days or hospital discharge, whichever came first
Arm/Group | Exparel Injectable Product | Bupivacaine Hydrochloride
All-Cause Mortality (participants affected / at risk) | 1/29 | 1/31
Serious Adverse Events (participants affected / at risk) | 5/29 | 5/31
Other Adverse Events (participants affected / at risk) | 3/29 | 5/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exparel Injectable Product (N=29) | Bupivacaine Hydrochloride (N=31)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 1
Pulmonary Arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension requiring aortic balloon pump (Cardiac disorders) | 0 | 1
Vasodilatory Shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exparel Injectable Product (N=29) | Bupivacaine Hydrochloride (N=31)
Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial Ectopy (Cardiac disorders) | 0 | 1
Hypoxia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT03270514/Prot_SAP_001.pdf